CLINICAL TRIAL: NCT01639222
Title: A Two Period, One-sequence Open-label Study of a Newly Developed Calcium Carbonate-vitamin D3 Chewable Tablet Formulation (Calcium 500 mg and Vitamin D3 800) Dosed for Three Days to Investigate the Effect on Urine Calcium and Serum Parathyroid Hormone (PTH) as Measurements of Intestinal Calcium Absorption in Healthy Postmenopausal Women and Healthy Men Compared to Baseline.
Brief Title: Human Pharmacology Trial of Calcium-vitamin D3 Tablet in Healthy Participants
Acronym: Osteopro
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CW-2200-401-RD; 2011-005786-21 (EudraCT Number); U1111-1124-2328 (Registry Identifier: WHO)
Record Dates: First submitted 2012-07-09; First posted 2012-07-12 (Estimated); Results first posted 2013-10-18 (Estimated); Last update posted 2013-10-18 (Estimated); Status verified 2013-08

CONDITIONS: Calcium Deficiency; Vitamin D Deficiency
Keywords: Drug therapy; Increase in calcium urinary excretion and PTH decrease in serum
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Calcium; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Calcium 500 mg and Vitamin D3 800 IU (Experimental): Period 1: Low calcium meals for up to 3 days.
  Period 2: Calcium 500 mg and Vitamin D3 800 IU chewable tablets, orally, once daily for up to 3 days with low calcium meals.
  Interventions: Drug: Calcium 500 mg and Vitamin D3 800 IU; Other: Low calcium meals

INTERVENTIONS:
Drug: Calcium 500 mg and Vitamin D3 800 IU — Calcium 500 mg and Vitamin D3 800 IU chewable tablets
  Other Names: Calcichew-D3 forte 500 mg/800 IU
Other: Low calcium meals — A normal Western European diet with reduced calcium content (400 mg per day).

SUMMARY:
The purpose of this study is to demonstrate that the intestinal absorption of calcium from a newly developed calcium carbonate-vitamin D3 chewable tablet formulation increases the amount of calcium excreted in urine and decreases parathyroid hormone (PTH) in serum as compared to baseline.

DETAILED DESCRIPTION:
The drug being tested in this study is called Calcichew. This study will look at calcium absorption in healthy postmenopausal women and healthy men.

The study will enroll approximately 55 healthy adults. All participants will receive Calcichew.

All participants will be asked to take one chewable tablet at the same time each day for three days in period 2 of the trial.

This trial will be conducted at one clinical site in Germany. The overall time to participate in this study is 4 weeks. Participants will make 9 visits to the clinic, and will be contacted by telephone 7days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy postmenopausal woman (last menses at least 2 years before signing informed consent and follicle stimulating hormone (FSH) confirming postmenopausal status) or a healthy male aged between 45 to 70 years inclusively
2. Was informed both verbally and in writing about the objectives of the clinical trial, the methods, the anticipated benefits and potential risks and the discomfort to which she/he might be exposed, and had given written consent to participation in the trial prior to any trial-related procedure
3. Is Caucasian
4. Is assessed as healthy based on physical examination, medical history, clinical laboratory, electrocardiogram (ECG), vital signs
5. Is a non-smoker (having abstained from smoking for at least 6 months)
6. Has a body mass index of 19 to 29.4 kg/m^2 (inclusively)

Exclusion Criteria:

1. Has a history of clinically significant allergies or idiosyncrasies to calcium or vitamin D3, or any inactive ingredient(s) of these products
2. Is a lactating or pregnant female participant
3. Female participants: Has a positive pregnancy test in serum at screening and in urine on Day -1 Period 1
4. Participant was previously enrolled into the current clinical trial
5. Has participated in the active treatment phase of another clinical trial where a persisting pharmacodynamic (PD) effect of the IMP of that clinical trial cannot be excluded (e.g. patient is well into a treatment free safety follow-up phase); or 10 times the pharmacokinetic (PK) half-life, whatever is longer but 30 days as minimum prior to the start of the clinical trial
6. Has been considered unable or unwilling to co-operate adequately, i.e. to follow clinical trial procedures and Investigator instructions adequately (e.g. language difficulties, etc.) or participant is anticipated not to be available for scheduled clinical trial visits/procedures
7. Has a dependency situation (e.g. person is kept in detention, Investigator in the current clinical trial, or a first-degree relative of a clinical trial Investigator, or is employee at the clinical trial site)
8. Has a hypersensitivity to soya or peanut
9. Abuse of alcohol or drugs
10. Has consumed ethanol within 48 hours prior to hospitalization verified by alcohol breath test (Alcotest®)
11. Has a history or current disease which might influence the trial objectives (e.g., urinary tract infection, urination problems [e.g., prostate hyperplasia] or urinary incontinence, renal insufficiency, nephrolithiasis, sarcoidosis, osteoporosis, calcium deficiency, hyper- or hypoparathyroidism, hypercalciuria, hypercalcaemia, calcium lithiasis, hyperphosphataemia, hypervitaminosis D, phenylketonuria, diabetes mellitus
12. Has creatinine clearance according to Modification of Diet in Renal Disease (MDRD) equation of < 60 mL/min
13. Has regular use of any medication. Treatment with biphosphonates in the past 5 years, amidorone in the past 6 months, calcium or fluoride supplements, diuretics, vitamin D preparations, estrogens or estrogen receptor modulators, enzyme inducing agents, teriparatide or parathyroid hormone (PTH(1-84)), bile sequestrants within 3 months before screening, and for all other drugs within 2 weeks before screening (or 6 times the half-life of the respective drug) whatever is longer
14. Has use of ultraviolet radiation cabins or sunbath longer than 1 h from 1 week before Day 1 of Period 1 until the End of Trial examination
15. Has an intake of milk and milk products, broccoli, dark-green vegetables, vegetables from the mustard green family, fatty fish, eggs, liver, and added salt within 7 days prior to hospitalisation
16. Has unusual diet habits and practicing vegetarians
17. Has beverages and food containing poppy seed (i.e. poppy seed rolls, poppy seed cake, milk shakes containing poppy seed) from 72 hours before drug screen to avoid interference
18. Has chinine, grapefruit- and star fruit-containing beverages and food, St. John's wort (known Cytochrome P450 (CYP450) inhibitors and inducers) within 7 days prior to hospitalization
19. Has excessive consumption of caffeinated beverages (more than five cups of coffee or equivalent per day)
20. Has consumption of xanthine-containing beverages and food (e.g. coffee, black and green tea, cola, chocolate) 48 hours prior to hospitalization
21. Has evidence of acute or chronic hepatitis B or C. Positive test for hepatitis B surface antigen (HBsAg), antibody to the hepatitis B core antigen (anti-HBc) or antibody to the hepatitis C virus (anti-HCV antibody), or human immunodeficiency virus (HIV) infection at screening
22. Has history of gastrointestinal surgery (except appendectomy) or any other gastrointestinal condition or disease that might influence (calcium) absorption
23. Has any condition, including laboratory findings or findings in the medical history or screening assessments that, in the opinion of the Investigator, constitutes a specific risk or a contraindication for the participant's participation in the trial or that could interfere with the trial objectives, conduct or evaluation
24. Has any comedication required during the trial.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Principal, Clinical Pharmacology, Study Director — Takeda
Locations (1):
- Mannheim, Baden-Wurttemberg, Germany

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Calcium 500 mg and Vitamin D3 800 IU
Started | 55
Completed | 55
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Calcium 500 mg and Vitamin D3 800 IU
Number analyzed (Participants) | 55
Age Continuous [Mean (Standard Deviation); unit: Years] | 57.07 (7.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 33
Region of Enrollment [Number; unit: Participants]
  Germany | 55
Height [Mean (Standard Deviation); unit: cm] | 172.71 (8.97)
Weight [Mean (Standard Deviation); unit: kg] | 77.28 (10.06)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 25.87 (2.33)
Creatinine Clearance [Mean (Standard Deviation); unit: mL/min/1.73 m²] | 86.60 (14.85)

OUTCOME MEASURES:

1. Primary Outcome: Amount of Calcium Excreted in Urine From 0 Hours up to 6 Hours Post Dose (Ca2+ Ae0-6h)
Description: Ca2+ Ae0-6h was calculated as the urine volume of the urine collected from 0 to 6 hours multiplied by the calcium concentration measured in urine.
Time Frame: Day 3 of Period 1 (Reference) and Day 3 in Period 2. Samples were taken 0-6 Hours post dose
Population: The Pharmacokinetic/Pharmacodynamic (PK/PD) Set included all enrolled subjects who received at least one dose of the mock treatment who had reliable values of either the primary PK parameter Ca2+ Ae0-6h in both periods or the primary PD parameter PTH AUC0-6h in both periods.
Measure: Mean (Standard Deviation); unit: mmol
Groups:
- Calcium 500 mg and Vitamin D3 800 IU: Period 2 (Days 4-6): Calcium 500 mg and Vitamin D3 800 IU chewable tablets, orally, once daily, followed by 200 mL of non-carbonated water, for up to 3 days with low calcium meals.
- Reference Treatment: Period 1 (Days 1-3): 200 mL of non-carbonated water (mock treatment) with low calcium meals for up to 3 days.
Arm/Group | Calcium 500 mg and Vitamin D3 800 IU | Reference Treatment
Number analyzed (Participants) | 55 | 55
mmol | 1.07 (0.49) | 0.63 (0.43)
Statistical Analysis 1: Comparison: Calcium 500 mg and Vitamin D3 800 IU vs Reference Treatment; The primary parameters were analysed in a mixed effects general linear model of the logtransformed values, including treatment as a fixed effect and subject as a random effect. The objective of the trial was met if the treatment contrast was statistically significantly different from 0 in the appropriate direction in a 2-sided test on a 5% significance level for both parameters. The 5% significance level for both primary parameters was not adjusted for multiple testing; Test type: Superiority or Other; Calcium-Vitamin D/Reference (%) = 179.72, 95% CI 2-sided [157.16 to 205.52] — Point estimates and 95% CIs for the treatment difference ratio (Calcium-Vitamin D/reference treatment) are provided on the original scale as a ratio * 100%

2. Primary Outcome: Area Under the Curve From 0 to 6 Hours Post Dose of Parathyroid Hormone (PTH AUC0-6h) in Serum
Description: The area under the curve from 0 to 6 hours post dose of parathyroid hormone (PTH AUC0-6h) in serum, calculated using the linear trapezoidal formula.
Time Frame: Day 3 in Period 1 (Reference) and Day 3 in Period 2. Samples were taken at predose, 0.5, 1, 2, 3, 4, and 6 hour post dose.
Population: PK/PD set
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | Calcium 500 mg and Vitamin D3 800 IU | Reference Treatment
Number analyzed (Participants) | 55 | 55
h*pg/mL | 202.02 (63.51) | 278.86 (79.71)
Statistical Analysis 1: Comparison: Calcium 500 mg and Vitamin D3 800 IU vs Reference Treatment; Test type: Superiority or Other; Calcium-Vitamin D/Reference (%) = 71.77, 95% CI 2-sided [68.83 to 74.84] — Point estimate and 95% CI for the treatment difference ratio (Calcium-Vitamin D /reference treatment) are provided on the original scale as a ratio * 100%

3. Secondary Outcome: Amount of Calcium Excreted in Urine From 0 to 6 Hours Post Dose Corected for Creatinine (Ae0-6h/Creatinine)
Description: To account for potential inaccuracies in urine collection, creatinine correction of calcium excretion was also assessed. Ca2+ Ae0-6h/Creatinine was obtained by dividing the urinary concentration of calcium by the urinary creatinine concentration.
Time Frame: Day 3 of Period 1 (Baseline) and Day 3 in Period 2. Samples will be taken 0-6 Hours postdose
Population: PK/PD set
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Calcium 500 mg and Vitamin D3 800 IU | Reference Treatment
Number analyzed (Participants) | 55 | 55
liters | 1.05 (0.92) | 0.69 (0.59)
Statistical Analysis 1: Comparison: Calcium 500 mg and Vitamin D3 800 IU; Test type: Superiority or Other; Calcium-Vitamin D/Reference (%) = 156.74, 95% CI 2-sided [121.66 to 201.93] — Point estimates and 95% CIs for the treatment difference ratio (Calcium-Vitamin D / reference treatment) are provided on the original scale as a ratio * 100%

ADVERSE EVENTS:
Time Frame: Up to 13 days.
Description: The investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. A safety follow-up phone call was conducted 7 to 12 days after last dosing.
Arm/Group | Calcium 500 mg and Vitamin D3 800 IU | Reference Treatment
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 5/55 | 6/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Calcium 500 mg and Vitamin D3 800 IU (N=55) | Reference Treatment (N=55)
Headache (Nervous system disorders) | 1 | 3
Dizziness (Nervous system disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Blood pressure increased (Investigations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights therefrom or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.